CLINICAL TRIAL: NCT00778843
Title: Efficacy and Safety of Viusid as Antioxidant and Immunomodulator Nutritional Supplement in Patients With Chronic Hepatitis C and Non-responders to Standard Antiviral Therapy. A Randomized and Double Blind Controlled Trial
Brief Title: Antioxidant and Immunomodulator Properties of Viusid in Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIU-CHC-08
Record Dates: First submitted 2008-10-21; First posted 2008-10-23 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; Oxidative stress; Antioxidant; Cytokines; Nutritional supplement
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Viusid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Viusid (Experimental)
  Interventions: Dietary Supplement: Viusid
- Placebo (Placebo Comparator): Placebo three oral sachets daily during 24 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Viusid — Viusid, three oral sachets daily during 24 weeks
  Arms: Viusid
Other: Placebo — Placebo three oral sachets daily during 24 weeks
  Arms: Placebo

SUMMARY:
The pathogenesis of chronic hepatitis C (CHC) is associated to severe oxidative stress and non-selective immunological disturbance that leads to necro-inflammation and progression of fibrosis. Previous trials suggested that antioxidant and inmunostimulant therapies may have a beneficial effect. The purpose of the study is to evaluate whether Viusid, a nutritional supplement with hepatoprotective properties, could ameliorate the oxidative stress and modulate the immune response in patients with CHC and non-responders to pegylated interferon plus ribavirin, during 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* HCV infection confirmed on a positive test for anti-HCV antibody and HCV RNA detectable in serum by Polymerase Chain Reaction.
* Histological diagnosis of chronic hepatitis.
* Patients who were non-responders to previous treatment with pegylated interferon and ribavirin or who had contraindicated the antiviral treatment.
* Age between 18 and 65 years.
* Ability to provide informed consent.
* Absence of significant alcohol ingestion (weekly ethanol consumption of less than 40 g)

Exclusion Criteria:

* Presence of other form of liver diseases (viral or autoimmune hepatitis, drug-induced liver disease, nonalcoholic steatohepatitis, metabolic and hereditary liver disease and α-1 antitrypsin deficiency).
* Pregnancy or lactation.
* Decompensated cirrhosis.
* Absence of clinical and ultrasonographic evidence of liver cancer, with α-fetoprotein levels ≤ 200 ng/ml.
* Refusal to participate in the study.
* Concomitant disease with reduced life expectancy.
* Severe psychiatric conditions.
* Drug dependence.
* Co-infection with hepatitis A or B or HIV.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The improvement of serum parameters related to oxidative stress (SOD, AT, MDA, MDA/HNE, GPx, GR, AOP, MPO, PAOP, GSH) at 24 weeks (end of the treatment). | 6 months
The improvement of serum parameters related to immune response (IFN alpha, IFN gamma, IL-1 alpha, IL-2, IL-6, IL-10, IL-12, TNF alpha, Anti TNF alpha, Cathepsin L) at 24 weeks (end of the treatment). | 6 months

SECONDARY OUTCOMES:
Improvement of aminotransferase levels (ALAT and ASAT) at 24 weeks (end of the treatment). | 6 months
Improvement of clinical symptoms and signs at 24 weeks (end of the treatment). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Vilar Gomez, Ph.D, Principal Investigator — National Institute of Gastroenterology
Locations (1):
- National Institute of Gastroenterology, Vedado, La Habana, Cuba

REFERENCES:
- [Result] Vilar Gomez E, Gra Oramas B, Soler E, Llanio Navarro R, Ruenes Domech C. Viusid, a nutritional supplement, in combination with interferon alpha-2b and ribavirin in patients with chronic hepatitis C. Liver Int. 2007 Mar;27(2):247-59. doi: 10.1111/j.1478-3231.2006.01411.x. PMID 17311621
- See also: Related Info — http://www.viusid.com